CLINICAL TRIAL: NCT00536861
Title: A Phase I Study of Radiotherapy Concurrent With Erlotinib (Tarceva®) in the Treatment of Brain Metastases From Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety Study of Radiotherapy and Concurrent Erlotinib (Tarceva®) for Brain Metastases From a Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Professor S Senan, VU Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUMC 2005/177
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-04

CONDITIONS: Non-Small Cell Lung Cancer; Brain Metastases
Keywords: erlotinib; cranial radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — Level 1 : erlotinib 100 mg/day from day -7 to the time of completion of 10 fractions of cranial irradiation, followed by 150 mg/day until disease progression or toxicity
  Level 2 : erlotinib 150 mg/day from day -7 before cranial irradiation, followed by 150 mg/day until disease progression or toxicity
  Other Names: Tarceva

SUMMARY:
Lung cancer is a leading cause of death worldwide. Brain metastases manifest as the first site of disease failure in between 15-30% of patients with non-small cell lung cancer (NSCLC). The standard treatment for patients with multiple brain metastases is whole brain radiotherapy but this results in only a modest survival of 3-6 months. Drugs that can enhance the effect of cranial irradiation (radiosensitizers) may improve the the response rates. Erlotinib (Tarceva) is an oral agent that has been registered for treatment in patients with metastatic NSCLC. Erlotinib has shown tumor activity in patients presenting with brain metastases, and preclinical studies show that it may be a radiosensitizer. As a prelude to studies investigating the combination of Erlotinib and cranial radiotherapy, the present study will be performed to evaluate the safety of combining both these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small cell lung cancer (NSCLC)
* Diagnosis of brain metastases on a contrast-enhanced CT scan or Gadolinium-enhanced MRI
* Patients who are not candidates for surgery or stereotactic radiosurgery
* RPA Class 1 or 2 (Karnofsky performance status > 70)
* Age > 18 years
* No previous radiotherapy, surgery or chemotherapy for brain metastases
* Patients must be able to take oral medication.
* Patients should not have any unstable systemic disease except lung cancer (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease).
* Granulocyte count > 1.5 x 109/L and platelet count > 100 x 109/L OK
* Serum bilirubin must be < 1.5 upper limit of normal (ULN).
* AST and/or ALT < 2 x ULN (or < 5 x ULN if clearly attributable to liver metastasis)
* Serum creatinine < 1.5 ULN or creatinine clearance > 60 ml/min
* Patients with reproductive potential must use effective contraception. For all females of childbearing potential a negative pregnancy test must be obtained within 72 hours before starting therapy.
* Able to comply with study and follow-up procedures
* Written informed consent.

Exclusion Criteria:

* Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, hepatic, renal or metabolic disease).
* Signs, symptoms or MRI findings consistent with leptomeningeal metastases.
* Concomitant use of phenytoin anticonvulsant medication
* Prior therapy with systemic anti-tumour therapy with HER1/EGFR inhibitors (as small molecule or monoclonal antibody therapy).
* Any other malignancies in the preceding 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Any significant ophthalmological abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating Oncologist and ophthalmologist.
* Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
* Nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To establish the safety of concurrent palliative whole brain radiotherapy and two doses of erlotinib in patients with brain metastases from NSCLC | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Senan, MD, PhD, Study Chair — Amsterdam UMC, location VUmc; Frank J Lagerwaard, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Egbert F Smit, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands